CLINICAL TRIAL: NCT02554019
Title: A Prospective, Double-blind, Randomized, Placebo-controlled, Repeated Dose, Multicentre Phase IIa Proof-of-Concept Study With BT063 in Subjects With Systemic Lupus Erythematosus
Brief Title: Proof-of-Concept Study With BT063 in Subjects With Systemic Lupus Erythematosus
Acronym: BT063 in SLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 990
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE, Lupus; IL10, IL-10, BT063, BT-063
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BT063 (Experimental): 50 mg BT063 administered by intravenous (IV) infusion 8 times
  Interventions: Biological: BT063
- Placebo (Placebo Comparator): Placebo administered by IV infusion 8 times
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BT063 — Repeated IV infusions over 12 weeks (at weeks 0, 1, 2, 4, 6, 8, 10, 12)
  Arms: BT063
Biological: Placebo — Repeated IV infusions over 12 weeks (at weeks 0, 1, 2, 4, 6, 8, 10, 12)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of repeated intravenous infusions of the study drug BT063 in patients with Systemic Lupus Erythematosus (SLE) compared with people who receive a placebo.

DETAILED DESCRIPTION:
Study 990 is a Phase IIa, proof-of-concept study of BT063 in subjects with SLE. This study is divided into 2 parts. After Part I an interim analysis will be performed. Each Part will enrol 18 subjects. Subjects will be randomly assigned to receive BT063 or Placebo 8 times over 12 weeks and will be followed for 4 months after their last dose.

ELIGIBILITY:
Inclusion Criteria:

* Eligible male and female subjects, Age ≥ 18 and ≤ 75 years with Body mass index ≥ 18 and ≤ 35 kg/m2 at screening visit
* Diagnosed SLE (defined by ≥ 4 of the 11 American College of Rheumatology (ACR) classification criteria for SLE) for at least 3 months before screening
* Moderate to severe SLE disease activity demonstrated by SLEDAI-2K total score ≥ 6, including skin and joint involvement
* CLASI Activity score ≥ 5 or at least 5 of 66/68 joints with pain and signs of inflammation
* Positive anti-nuclear antibodies (ANA) test at screening
* No change in concomitant medication for SLE activity maintenance and symptom control regarding type of medication and dose level for at least 8 weeks prior to baseline (for steroids and NSAIDs/pain medication 2 weeks)
* Normal electrocardiogram (ECG)

Exclusion Criteria:

* Active, severe neuropsychiatric SLE defined as any neuropsychiatric element scoring BILAG level A disease or lupus nephritis
* Diagnosed psoriasis
* Presence or history of malignancy within the previous 5 years
* Systemic antibiotic treatment within 2 weeks before baseline visit
* A positive diagnosis for viral hepatitis B or hepatitis C or Human immunodeficiency virus (HIV) or tested positive for tuberculosis as assessed or recent infection with Herpes Zoster or Herpes Simplex (Type 1 and Type 2), Epstein-Barr virus (EBV) or cytomegalovirus (CMV) infection or reactivation at screening
* Clinically significant hematologic abnormalities attributed to SLE: Haemoglobin < 8 g/dL; Platelets < 50 E9/L; Leucocytes < 2.0 E9/L
* Active or history of inflammatory bowel disease (including active or history of colitis)
* Received the following medications: - Rituximab within the last 48 weeks before screening - Belimumab within the last 12 weeks before screening - IV immunoglobulin (Ig) within the last 12 weeks before screening - Intramuscular (IM) or intra-articular glucocorticosteroids within the last 4 weeks before screening - IV cyclophosphamide within the last 6 months before screening - IV glucocorticosteroids (pulse therapy) within the last 6 months before screening
* Pregnant or nursing women or women who intend to become pregnant
* Known intolerance to immunoglobulins or comparable substances (e.g., significant vaccination reaction)
* Known intolerance to proteins of human origin
* History of clinically significant drug or alcohol abuse within the last 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nemanja Damjanov, Professor, Principal Investigator — Institute of Rheumatology, University of Belgrade School of Medicine
Locations (14):
- Belarus (5):
  - Study Site 37505, Homyel
  - Study Site 37501, Minsk
  - Study Site 37502, Minsk
  - Study Site 37503, Minsk District
  - Study Site 37504, Vitebsk
- Georgia (2):
  - Study Site 99501, Tbilisi
  - Study Site 99502, Tbilisi
- Poland (4):
  - Study Site 48003, Bialystok
  - Study Site 48004, Krakow
  - Study Site 48002, Poznan
  - Study Site 48001, Warsaw
- Serbia (3):
  - Study Site 38101, Belgrade
  - Study Site 38103, Belgrade
  - Study Site 38102, Niška Banja

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 36 subjects were enrolled in study parts I and II (18 in part I and 18 in part II). 12 subjects in part I received 50 mg BT063, 12 subjects in part II received 100 mg BT063. 6 subjects in part I and 6 subjects in part II received Placebo and were pooled for analysis. Only final results and no partial or interim results are presented.
Groups:
- BT063 50 mg: 50 mg BT063 administered by intravenous (IV) infusion 8 times
  BT063: Repeated IV infusions over 12 weeks (at weeks 0, 1, 2, 4, 6, 8, 10, 12)
- BT063 100 mg: 100 mg BT063 administered by intravenous (IV) infusion 8 times
  BT063: Repeated IV infusions over 12 weeks (at weeks 0, 1, 2, 4, 6, 8, 10, 12)
Period: Overall Study
Arm/Group | BT063 50 mg | BT063 100 mg | Placebo
Started | 12 | 12 | 12
Completed | 10 | 12 | 10
Not Completed | 2 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BT063 50 mg | BT063 100 mg | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.77) | 50.7 (7.18) | 48.6 (13.5) | 45.6 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 12 | 33
  Male | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 12 | 12 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events (Including SAEs and AEs leading to discontinuation) from Baseline through End of Trial Visit (Week 14)
Time Frame: Baseline through End of Trial Visit (Week 14)
Measure: Count of Participants; unit: Participants
Arm/Group | BT063 50 mg | BT063 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Subjects with TEAEs | 5 | 8 | 8
  Subjects with TEAEs leading to early termination | 1 | 0 | 0
  Subjects with treatment-emergent SAEs | 1 | 1 | 0
  Subjects with drug-related TEAEs | 1 | 2 | 0
  Subjects with severe TEAEs | 0 | 0 | 0
  Subjects with TEAEs leading to death | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Changes of Safety Parameters
Description: Number of Participants with changes in vital signs, ECGs, Safety laboratory parameters (full blood count including white differential count, clinical chemistry, thyroid hormones, urinalysis, and faecal occult blood test), Development of anti-drug antibodies against BT063 (anti-BT063), Immunological status of potential viral and bacterial infections (HBV, HCV, HIV, tetanus, diphtheria tuberculosis), EBV / CMV Serology, Premature withdrawals.
Time Frame: Baseline through End of Trial Visit (Week 14)
Measure: Count of Participants; unit: Participants
Arm/Group | BT063 50 mg | BT063 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Improvements of Joints
Description: Number of Participants with 50% improvement of swollen/tender joints. A total of 66/68 joints was assessed for the swollen/tender joint count. A joint that is normal (no tenderness or swelling), without signs of inflammation will be graded as 0. A joint with tenderness will be graded as 1 for tender joint count and a joint with swelling will be graded as 1 for swollen joint count. Joints suspected or known to have ischemic osteonecrosis are not to be taken into consideration. Higher scores indicate more disease activity.
Time Frame: At week14 and week 28
Population: Intension-To-Treat Set included 36 subjects (12 of each Group). At week 14, 1 subject in Placebo Group had no end of Treatment result; at week 28, 1 subject of 50 mg and 2 subjects of Placebo had no results. The efficacy outcome was based on observed cases.
Measure: Count of Participants; unit: Participants
Arm/Group | BT063 50 mg | BT063 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants
  50% improvement in swollen joints at week 14: number analyzed (Participants) | 12 | 12 | 11
  50% improvement in swollen joints at week 14 | 8 | 5 | 8
  50% improvement in swollen joints at week 28: number analyzed (Participants) | 11 | 12 | 10
  50% improvement in swollen joints at week 28 | 7 | 4 | 7
  50% improvement in tender joints at week 14: number analyzed (Participants) | 12 | 12 | 11
  50% improvement in tender joints at week 14 | 5 | 7 | 6
  50% improvement in tender joints at week 28: number analyzed (Participants) | 11 | 12 | 10
  50% improvement in tender joints at week 28 | 7 | 6 | 6

4. Secondary Outcome: Number of Participants With Improvement of Skin
Description: Number of Participants with 50% improvement in Cutaneous Lupus Erythematosus Disease Area and Sensitivity Index (CLASI) Activity score. The CLASI is an assessment over 13 body regions (scalp, ears, nose - including malar area, rest of the face, V-area neck - frontal, post. neck & shoulders, chest, abdomen, back and buttocks, arms, hands, legs, feet) and consists of 2 scores: total activity score and total damage score. Only the activity score was used in this study.
  The minimum score possible on this scale is 0 and the maximum score is 70. The higher scores mean a worse outcome.
Time Frame: At week14 and week 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BT063 50 mg | BT063 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants
  50% improvement in CLASI Activity score at week 14: number analyzed (Participants) | 12 | 12 | 11
  50% improvement in CLASI Activity score at week 14 | 6 | 5 | 3
  50% improvement in CLASI Activity score at week 28: number analyzed (Participants) | 11 | 12 | 10
  50% improvement in CLASI Activity score at week 28 | 7 | 4 | 3

5. Secondary Outcome: Percent Changes in Systemic Lupus Erythematosus Disease Activity Index 2000
Description: Percent changes in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) scores from baseline SLEDAI-2K score.
  The SLEDAI-2K is a global index that measures SLE disease activity. It includes 24 items for the 9 organs/systems. Scores range from 0 to 105; a score of 6 is considered clinically important. The index measures disease activity within the last 10 days. Higher scores mean worse outcome. Negative percent change means reduced disease activity.
Time Frame: Baseline to week 14 and at week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | BT063 50 mg | BT063 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
percentage of change
  Percent changes in SLEDAI-2K scores at week 14: number analyzed (Participants) | 12 | 12 | 11
  Percent changes in SLEDAI-2K scores at week 14 | -29.3 (31.43) | -18.0 (37.304) | -18.2 (25.75)
  Percent changes in SLEDAI-2K scores at week 28: number analyzed (Participants) | 11 | 12 | 10
  Percent changes in SLEDAI-2K scores at week 28 | -28.9 (36.05) | -24.4 (35.19) | -13.5 (32.36)

ADVERSE EVENTS:
Time Frame: Incidence of AEs (including SAEs and AEs leading to discontinuation) from baseline through End of Trial Visit (Week 14)
Arm/Group | BT063 50 mg | BT063 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 6/12 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT063 50 mg (N=12) | BT063 100 mg (N=12) | Placebo (N=12)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — mild; not related; recovered
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — moderate; not related; recovered
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — moderate; not related; recovered
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT063 50 mg (N=12) | BT063 100 mg (N=12) | Placebo (N=12)
ASTHENIA (General disorders) | 0 (0) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall not publish, present, or use any Study data or results arising out of the performance of the Study for their own instruction, research, or publication purposes without the prior express written consent of Sponsor, which consent may be withheld at Sponsor's discretion.

DOCUMENTS (2):
  • Study Protocol (2015-03-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT02554019/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT02554019/SAP_001.pdf